# Protocol Title: Telehealth Delivery of Treatment for Sleep Disturbances in Young Children with Autism Spectrum Disorder

Funding: Department of Defense

Principal Investigator: Cynthia Johnson, PhD

#### **Background**

#### ASD is a Major Health Problem in Need of Evidenced-Based Treatments.

Current estimates of the prevalence of ASD range from 6.2 to 14.7 per 1000.<sup>1,2</sup> In addition to the core features of ASD (social communication deficits; repetitive and restrictive behaviors), as many as 70% of children with ASD have additional problems such as hyperactivity, disruptive behavior, and anxiety severe enough to warrant treatment.<sup>3-8</sup> An estimated 44 to 80% of children with ASD also have sleep disturbances.<sup>9-12</sup> This wide range reflects differences in the source of sample, assessment methods and severity level (mild to severe). The estimate of 80% likely includes children with mild sleep disturbance. Children with ASD and moderate or greater levels of severity require intervention.<sup>13</sup> Providing appropriate treatment for children with ASD is a challenge to the service system, with current costs estimated to be \$125 billion annually.<sup>14</sup> Treatment approaches commonly used for core and associated features include behavior therapy,<sup>15-17</sup> comprehensive educational interventions<sup>18,19</sup> and pharmacotherapy.<sup>20,21</sup> The heightened recognition and increased demand for services, however, occurs against a backdrop of insufficient evidence for many treatments.<sup>22-25</sup> There is a pressing need to conduct well-designed studies to expand the portfolio of *empirically supported*, *time-limited and cost-effective interventions* to meet rising demand and guide clinical practice.<sup>26</sup>

According to the World Health Organization, a major obstacle for access to adequate services for children with disabilities is the lack of trained specialists.<sup>27</sup> Although children with ASD account for 10–14% of those referred for mental health treatment, only 5% of mental health practitioners consider themselves prepared to treat children with ASD.<sup>28</sup> Moreover, training in behavioral health programs on the assessment and treatment of pediatric sleep disturbances is limited.<sup>29</sup> As a result, the demand for treatment of children with ASD and sleep disturbances far outpaces the availability of empirically supported interventions and skilled providers in the community. This lack of access often results in long waiting lists for services and families resorting to treatments without empirical support.<sup>30</sup> In a randomized trial of 180 young children with ASD, we showed that parent training was superior to parent education for reducing disruptive behavior.<sup>31</sup> This project will test whether telehealth delivered parent training for sleep problems is superior to parent education in children with ASD.

#### Importance of Sleep.

Biological and environmental factors play a role in the development and maintenance/disruption of the sleep-wake cycle. The hypothalamus controls the timing of sleep, body temperature and cortisol production. Melatonin (produced by the pineal gland) affects sleep-wake patterns via feedback between the pineal gland and hypothalamus. This hormone is suppressed by exposure to bright light. Factors such as light perception, social cues, ambient temperature, noise levels, and internal body signals (hunger, body temperature) also contribute to the sleep-wake rhythm. Sleep requirements vary by age: children 2 to 5 years require 11-13 hours of sleep per day; school-age children require 10-11 hours. 33-37

Over fifty years of research attest to the critical need for adequate sleep. Sleep plays a central role in early brain maturation <sup>38-40</sup> and plasticity. <sup>41-47</sup> Inadequate sleep in school-age children can impair cognitive functions such as working memory and abstract thinking, <sup>48-51</sup> motor reaction time; <sup>52</sup> attention, <sup>45,48,51,53-59</sup> emotion regulation <sup>48,51,60-62</sup> and academic functioning. <sup>54,57,63,64</sup> Although limited, available evidence suggests a clear link between disrupted sleep and daytime behavior problems in young children. <sup>62,63,65</sup> Sleep disturbances in young children may also have adverse effects on family functioning due to parental sleep deprivation. <sup>66-68</sup>

#### Sleep, Mental Health & Physical Health.

Sleep disturbances are associated with several mental health disorders including anxiety, depression, attention deficit hyperactivity disorder (ADHD), post-traumatic stress, and bipolar disorder. Several studies show the common co-occurrence of sleep problems and emotional problems in children. Heart Emerging data link sleep disruption to the *onset* of internalizing and externalizing problems in children. These findings have prompted a shift in treatment paradigms to address sleep difficulties alongside the emotional and behavioral problems or even as a first step in the treatment plan. Moreover, there are physical health implications for Version 1.2: 7-12-2018

chronic, inadequate sleep and poor sleep quality.<sup>83-85</sup> Collectively, there is compelling evidence that intervening early on sleep disturbances in young children with ASD could offset a range of untoward events and maximize a child's participation in early therapeutic and educational activities.

#### Sleep Disturbances in Children with ASD.

The prevalence of sleep problems in the general pediatric population is estimated at 25%. <sup>86</sup> By contrast, poorly regulated sleep patterns (trouble falling asleep, mid-sleep awakening and early morning awakening) affect as many as 80% of children with ASD regardless of cognitive functioning level. <sup>10,11,67,87-98</sup> Although severity of sleep dysregulation in children with ASD varies from mild to severe, children with moderate or greater sleep problems require treatment to avert the associated adverse effects of inadequate sleep. Closely related problems for children with ASD include noncompliance with bedtime routines, difficulty establishing essential elements of sleep hygiene due to over-arousal and sleep-onset association problems (e.g., only able to fall asleep somewhere other than bed, requires certain objects or person to be present for sleep onset), <sup>12</sup> resulting in overall lower sleep quality. <sup>99</sup>

Johnson<sup>10</sup> long ago proposed that the core social communication deficits of ASD, and often co-occurring cognitive deficits, interfere with the child's capacity for self-soothing. Consequently, children with ASD may be less able to promote *sleep onset* independently or return to sleep upon waking after sleep onset.<sup>10</sup> Children with ASD may also have difficulty understanding social and environmental cues that are part of the *bedtime routine*. Some children with ASD develop idiosyncratic bedtime routines that hinder sleep such as insisting on toys be arranged just so with attendant disruptive behavior that interferes with settling down.<sup>99</sup> Co-occurring gastrointestinal problems, seizures, anxiety, depression, ADHD, or medication side-effects (e.g., stimulants, serotonin reuptake inhibitors) may also interfere with sleep patterns.<sup>90,100-106</sup> Alteration in melatonin secretion in children with ASD may contribute to sleep disturbance.<sup>107,108</sup> Several studies have reported markedly lower mean plasma melatonin levels and lower urinary excretion of melatonin sulfate (MEL-S, also known as 6-MEL-S) in ASD compared to typically developing controls.<sup>109-111</sup> In sum, disruptive behavior, elaborate bedtime routines, poor self-soothing and understanding of environmental cues, neurochemical alterations, and concurrent medical problems may interfere with developing a stable sleep-wake cycle in children with ASD.

Disordered sleep in children with ASD can amplify already delayed social interactions, repetitive behaviors, affective problems, inattention/hyperactivity, and irritability. 88,112-117 Given the documented detrimental effects of sleep disturbance on cognition, attention, memory consolidation, and daytime behavioral adjustment, addressing sleep disturbances in young children with ASD may promote overall improvement and fuller use of educational and therapeutic interventions. Sleep difficulties in children with ASD produce significant stress on caregivers and negative attitudes toward the child. 88,118-120 Parents of children with ASD have poorer sleep quality than parents of typically developing children. 121,122 Sleep problems in the child may contribute to lower quality of sleep in mothers, 123 and are inversely correlated with maternal depressive symptoms. 124 Interventions that improve sleep in the child may reduce parental stress and improve mood and overall health.

#### Interventions for Sleep Disturbance in Children with ASD.

Supplemental melatonin, which is safe and inexpensive, has shown promise as a treatment for sleep onset delay in children with ASD.<sup>32,109,125-133</sup> However, melatonin does not address behavioral bedtime resistance, teach self-soothing to promote sleep, and may not be helpful for night wakings.<sup>109,133</sup> Not surprisingly, behavioral interventions for sleep disturbances remain first line treatments for insomnia in general pediatrics.<sup>134,135</sup> However, behavioral interventions for sleep disturbances in children with ASD have not been carefully studied. Ironically, surveys indicate that most parents of children with ASD favor behavioral approaches over sleep-enhancing medications.<sup>120</sup> Based on successful behavioral interventions for sleep onset and maintenance problems used in typically developing children, similar approaches have been used clinically in children with ASD with some success.<sup>96,135</sup> Specific adaptations for children with ASD and other developmental disorders include establishment of routines, environmental modifications, placing sleep restrictions on the child, extinction procedures, and scheduled awakenings.<sup>136-146</sup> The time is right to pursue a well designed randomized trial targeting sleep disturbances in children with ASD to guide clinical practice with the goal of optimizing the reach of the intervention via telehealth.

#### **Behavioral Parent Training in ASD.**

Parents confront daily struggles in rearing a child with ASD. Sleep disturbances present yet another challenge. Parent training (PT) is a fitting treatment model for sleep problems in young children with ASD for several reasons: 1) the central role of parents in promoting the development of children with ASD; 2) the demonstrated feasibility of parent training in the treatment of sleep problems (see below); and 3) the negative impact of sleep disturbances on the child and family. To date, structured PT interventions have focused largely on child language, adaptive skills, joint attention and other social communication behaviors. There is a growing body of empirical support for the efficacy of PT in children with ASD and disruptive behavior. In two previous large-scale multi-site trials, we showed that PT was effective for reducing disruptive behavioral problems and improving daily living skills compared to parent education. Our PT program included one session on sleep problems, which was helpful for some children. For children with ASD and moderate to severe sleep problems, however, more intensive and focused treatment on sleep may be required.

In a review of 24 published studies on behavioral interventions that targeted sleep problems in children with ASD and other developmental disabilities, most studies were small case series or single subject design studies. These studies set the stage for a large RCT as the next step in keeping with the recommendations of an NIMH convened workgroup. 155 To date, there have been only two large-scale RCTs of a behavioral intervention for sleep disturbances in children with ASD. 143 Cortesi and colleagues 156 compared the efficacy of 4 sessions of PT to PT plus melatonin (MLT), MLT alone and placebo in a sample of 160 4-10 year-olds with ASD. After 12 weeks, all three active treatments showed superiority to placebo in sleep onset latency (SOL) and wakings after sleep onset on actigraphy and a parent completed questionnaire. There was a statistical trend favoring combined treatment. In a randomized sample of 80 children with ASD, ages 2-10 years with sleep onset problems, Malow and colleagues compared a single parent individual educational session to two group sessions. Both programs showed improvement in SOL and modest improvement in sleep efficiency on actigraph. <sup>157</sup> Although these studies expand the evidence-base on sleep interventions for children with ASD, both have notable limitations. The four-group study by Cortesi et al. 156 excluded children with behavioral problems, which limits generalizability. In addition, subjects whose treatment compliance fell below 80% (n=16) were excluded from the analysis. The Malow et al. study was brief and focused primarily on sleep latency. These studies were all delivered in a tertiary clinical setting. These settings are limited to their access to families who may have to travel distances and may have long waiting lists.

Although prior research documents the high rate of moderate or greater sleep problems in children with ASD and the potentially detrimental effects, available evidence on intervention is encouraging but inconclusive. The time is right for an innovative telehealth trial of an exportable parent training intervention for sleep disturbances in young children with ASD. In a prior pilot study (R34MH082882 – PI Johnson<sup>97</sup>), we showed that our SPT for young children with ASD and sleep disturbances was acceptable to parents and reliably delivered by therapists (see Support section for reference of the published paper of this pilot trial). We now propose a RCT to test the efficacy of telehealth delivered SPT against parent education – which will control for time and attention.

#### Telehealth and ASD

Telehealth, also referred to as telemedicine and more recently telepractice, is the use of communication technologies to allow delivery of services across a range of conditions and over geographical distances. The capacity of telehealth to deliver empirically based interventions for children with ASD holds promise as a means to close the gap between demand for services and the availability of autism specialist in underserved and rural areas such as those making up large swaths of the state of Florida. Despite the potential for telehealth in the delivery of assessment and treatment of children with ASD, this has received limited research attention. A few studies have demonstrated the use of telehealth to delivery interventions that are acceptable to parents but this is a under developed area at present. Treatment for sleep is particularly suited for telehealth as this allows for more ecologically sound delivery of the intervention close to bedtime.

#### **Preliminary Data**

#### Do previous findings suggest SPT for sleep disturbances in children ASD can be effective?

In our prior NIH-funded pilot study (R34MH082882; Johnson, Turner, Foldes, Brooks, Kronk, Wiggs <sup>97</sup>), we showed that our structured 5 session parent training intervention for young children with ASD and sleep disturbances was acceptable to parents and reliably delivered by therapists in a clinic setting. Parents attended 97% of expected sessions; parent satisfaction was high. Treatment fidelity (therapist integrity and parent

Figure 1. Mean CSI Scores with Effect Sizes



adherence) was over 95%. The SPT group improved significantly more than the comparison group based on the primary outcome of the CSI of the MSPSQ (see Figure 2). Using a benchmark of ≥30% improvement on the CSI, the SPT group had a positive response rate of 60% compared to the PE group (33%). Again, this study was delivered in a tertiary, specialized setting requiring parents to make many trips to an urban area; some families traveled over two hours to participate.

#### What was learned from our previous study?

A number of lessons were learned from this earlier study which will benefit this current project. First, telehealth SPT will be delivered over 10 weeks (versus 8 weeks in the previous study). This provides more time for parental application of strategies in the home and more time to detect change. Second, the time and distance was a barrier for potential participants who would have otherwise met eligibility criteria.

#### What is the impact of child sleep disturbance on parents?

In 49 children (mean =  $3.48\pm1.02$  years) with ASD and their parents, the CSI was highly correlated with a measure of parent sleep quality (Pittsburgh Sleep Quality Index) (r=.52; p <.001). As sleep disturbances in children increased, parents' sleep worsened. 164

#### **Experience with the use of telehealth platforms?**

Dr. Johnson and colleagues are currently conducting an NIH-funded multi-site pilot study of a behaviorally-based parent training program targeting <u>feeding problems</u> in young children with ASD. The study utilizes a HIPAA-compliant teleconferencing system (VSEE) to provide clinic-to-home parent-child coaching during mealtimes even though the parent training sessions per se are provided in a clinic setting. All families randomized to treatment thus far (N=22) have been able to successfully connect through the system in order to receive in-vivo coaching from a therapist during mealtimes. In conducting this trial, the idea to use a telehealth platform in the delivery of SPT was generated. The use of a telehealth platform has particular advantages to address sleep disturbances. Aside from the advantage of reaching families who may be a distance from a university setting, the use of the platform allows more flexibility in scheduling to include scheduling in the evening around bedtime, allows for real-time parent-child coaching soon after learning about the procedures discussed, and overall greatly enhances the ecological validity of the intervention.

For this trial, the telehealth platform will be the Cleveland Clinic Express Care Online. This platform is also HIPAA-compliant, and has capabilities that are similar to VSEE.

# **Objectives / Specific Aims / Hypotheses**

Across a range from mild to severe, as many as 80% of children with autism spectrum disorder (ASD) have sleep disturbances. 9,12,94,97,165 Sleep problems in typically developing children have adverse impacts on daytime behavior, emotion regulation, learning, physical health, as well as parent and family functioning. 52,84,123,166,167 For children with ASD whose development is compromised by a range of deficits, the impact of sleep disturbances may be more far reaching. Given the improved recognition of ASD and the prevalence of sleep disturbances in this pediatric population, increased demand for treatment of children with ASD and sleep disturbances in pediatric sleep clinics, community behavioral health clinics and specialized ASD programs is inevitable. Accumulating data indicate that behaviorally based interventions for sleep disturbance can be effective. Despite the recommendation for these interventions in pediatrics broadly 168 and ASD specifically, there have been few randomized controlled trials of behavioral interventions for sleep disturbance in children with ASD and none of these small trials included telehealth.

In response to FY17 ARP Clinical Trial Award funding opportunity (W81XWH-17-ARP-CTA), this four-year study will test the efficacy of a behavioral parent training intervention specifically designed for sleep disturbances and delivered individually through the HIPAA compliant Cleveland Clinic Express Care Online telehealth platform. This study will address the following areas of interest: 1) Behavioral, cognitive and other non-pharmacological therapies and 2) Therapies to alleviate conditions co-occurring in ASD (e.g, sleep disturbances).

A sample of 90 children with ASD (ages 2 to less than 7 years) and moderate or greater sleep disturbances will be **randomly** assigned to 10 weeks of a structured, 5 session sleep parent training (SPT) program or 10 weeks of a structured, 5 session parent education (SPE) program. Our recently completed randomized pilot trial (n=33) demonstrated that SPT is acceptable to parents and provided promising preliminary efficacy data. We now propose an efficacy study of SPT delivered individually via telehealth platform for sleep disturbances in young children with ASD. We will also examine the impact of SPT on the child's overall functioning and parental quality of life. Children who do not show a positive response to SPE will be offered SPT at no charge by study therapists.

#### **Primary Aim**

To evaluate the efficacy of telehealth deliver of SPT (n=45) compared to telehealth delivery of SPE (n=45) for sleep disturbance in children with ASD.

<u>Hypothesis 1</u>: After 10 weeks of treatment, children whose parents receive SPT will show greater improvement in sleep as evidenced by reduction on the Composite Sleep Index (CSI) of the modified Simonds and Parraga Sleep Questionnaire<sup>97,144</sup> compared to children whose parents receive SPE.

<u>Hypothesis 2</u>: After 10 weeks of treatment, children whose parents receive SPT will show a significantly higher rate of overall improvement on the Improvement scale of the Clinical Global Impression (CGI-I), as assessed by an independent evaluator masked to group assignment, compared to children whose parents receive SPE. Ratings of Much Improved or Very Much Improved will be used to define positive response.

<u>Hypothesis 3</u>: After 10 weeks of treatment, children whose parents receive SPT will show significantly reduced disruptive behavior on the parent-rated Irritability subscale of the Aberrant Behavior Checklist (ABC) compared to children whose parents receive SPE.

<u>Hypothesis 4</u>: At post-treatment follow up on Week 16, children in the SPT group will continue to show significantly lower scores on the CSI and a significantly higher rate of positive response on the CGI-I scored by an Independent Evaluator masked to treatment assignment compared to children in SPE.

#### **Secondary Aim**

To evaluate the impact of SPT on parental quality of life (parental stress, parental competency, mental health and sleep quality) compared to SPE.

<u>Hypothesis 1</u>: After 10 weeks of treatment, parents enrolled in SPT will report lower levels of stress and higher levels of competency and health as measured by the Parenting Stress Index (PSI), Parenting Sense of Competence (PSOC), and Parent Health Questionnaire (PHQ) compared to parents in SPE. <u>Hypothesis 2</u>: After 10 weeks of treatment, parents receiving SPT will report improved sleep for themselves on the Pittsburgh Sleep Quality Index (PSQI) compared to parents receiving SPE.

#### **Study Design**

As shown in Figure 2, 90 eligible subjects will be randomly assigned in a 1:1 ratio to sleep parent training (SPT) or sleep parent education (SPE) using a randomized block design (random blocks of sizes 4 and 8), with allocation concealed to investigators. Both treatments provide 5 individually-delivered sessions over 10 weeks. All participants will be assessed on study outcomes at Weeks 5 and 10 as well as 6 weeks post-treatment. *Parents who complete SPE may receive SPT after the Week 16 evaluation*.

#### **Inclusion/Exclusion Criteria**

#### Inclusion Criteria

- 1. Both genders  $\geq 2$  and  $\leq 7$  years of age [RATIONALE: Based on pilot findings with similar age range  $^{97}$ ]
- 2. Clinical diagnosis of ASD corroborated by the Modified Checklist for Autism in Toddlers<sup>169</sup> or the Social Communication Questionnaire.<sup>170</sup> We will collect the MCHAT on children 2-3 years of age, both MCHAT and SCQ on children >3-<6, and SCQ for children >6-7 years of age via REDCap (Research Electronic Data Capture,<sup>171</sup> see details in the Data Management section). We will use recommended cutoff scores (score of 8 for MCHAT and 15 for SCQ) for inclusion.
- 3. Score of  $\geq 5$  on the CSI and a Clinical Global Impression Severity (CGI-S) score of Moderate or greater. [RATIONALE: This CSI score reflects moderate sleep disturbances and was the entry score in prior studies by

Johnson et al<sup>97</sup> and Wiggs and Stores;<sup>144</sup> The CGI-S score of Moderate is commonly used as clinician validation of parent ratings.]

4. Medication and supplement free or on stable medication or supplements (no changes in the past 6 weeks and no planned changes for 16 weeks). [RATIONALE: Many children with ASD are on medication for various target behaviors that may affect sleep. Children on stable medication (or supplement) for sleep, who otherwise meet study entry criteria, will be included because residual sleep problems remain. Including children on stable medication (or supplement) will enhance the representativeness of the study sample.]

Figure 2



5. Parental proficiency in spoken and written English language. [RATIONALE: At the

written English language. [RATIONALE: At the present time, study materials and many of the study measures are available only in English. If SPT is efficacious, we will take the next steps to translate the manual]. *Exclusion Criteria* 

- 1. Children with a serious medical condition or a known or suspected medical cause for sleep disturbances (e.g., nocturnal seizures, unresolved gastrointestinal problems such as reflux or constipation).
- 2. Children with a psychiatric disorder or serious behavioral problems requiring immediate treatment.


3. Children with known or suspected sleep apnea, restless legs, or periodic limb movements during sleep, or a circadian-based sleep disorder (e.g. delayed or advanced sleep phase syndrome) based on history and all available information. [RATIONALE: Children with these conditions warrant a different treatment. We will provide referrals as needed.]

#### Recruitment

To randomize 90 subjects, we expect to screen approximately 120 subjects. Approved advertisements about the project will be circulated within the Cleveland Clinic Center for Autism and other key programs within the Cleveland Clinic systems. Regional autism programs in the community will also be approached and provided information about the study. In the state of Florida, the university-based Centers for Autism and Related Disabilities (CARDS), with whom the PI has relationships, have over 3000 children registered in this young age range. The study will also be posted on ClinicalTrials.com. With distance not a limiting factor with telehealth delivery, recruitment is anticipated to be easily attainable.

# **Study Procedures and Randomization Visit Schedule for Assessments**

#### Screening Visit:

Subjects who appear to be eligible on a telephone interview will be scheduled for an Express Care Online screening visit. After obtaining informed consent which the family will access and sign using a REDCap link, parents will completed the assessment measures to confirm eligibility (see Table 1).

#### Baseline Visit:

Once eligibility is confirmed, an Express Care Online baseline visit will occur within 7-14 days of screening to complete additional measures (see Table 1). Parents will also be instructed to take photographs of their child's sleep environment for review and treatment planning during the baseline visit.

#### Randomization:

Participants will be randomly assigned to SPT or SPE at the conclusion of the baseline visit in a 1:1 ratio. A randomized block design (with random blocks of size 4 and 8) will be used to ensure balance as well as maintaining the blinding of allocation assignment by investigators. The randomization module in REDCap will be utilized to reveal the assignment for each participant. Assignment status will be maintained in a separate REDCap data set, with a shared identifier to be able to link to the study database for final analysis. Limited study staff who are not masked to treatment group assignment will have access to this database.

#### Post-randomization Assessments:

Assessments for both groups will be repeated at Weeks 5, 10 and 16 (see Table 1). The classification of positive or negative response will be made at Week 10 (endpoint of the randomized trial). To protect the treatment blind for IEs and to assess the effects of time within each treatment, all subjects will be asked to return at Week 16.

# **Establishing Study Inclusion Criteria, & Subject Characterization**

#### Developmental, Medical, & Sleep History.

This questionnaire will be completed by the parent / caregiver at screening to document prenatal, perinatal or postnatal medical and developmental histories including, sleep, medication and past assessments (see Survey and Questionnaires section). If any questions arise that would exclude the child and/or warrant other care, we will discuss with the family. This history form requires 20-30 minutes to complete.

The Modified Checklist for Autism in Toddlers (M-CHAT-R)<sup>169</sup> is a 20 items screening measure to detect high risk toddlers for ASD. This measure has been well validated and widely used. Scores between 8-20 are in the high risk range. We will use a score of ≥8 to corroborate the clinical diagnosis required for CARD registration. Internal consistency across all of the M-CHAT-R items fell below the adequate threshold (Cronbach's alpha = 0.63); however, when the second stage of the M-CHAT-R was examined internal consistency was found to be adequate (Cronbach's alpha = 0.79). The M-CHAT-R initial scoring, with a cutoff score of 3, has a sensitivity of 0.911, and specificity of 0.955, both with a 95% CI. <sup>169</sup> M-CHAT requires 10-15 minutes to complete and is written on 4<sup>th</sup> grade reading level.

The <u>Social Communication Questionnaire</u> (SCQ)<sup>170</sup> is a parent report screening measure for autism spectrum Version 1.2: 7-12-2018

Page **8** of **27** 

disorders (ASD) based on the Autism Diagnostic Interview-Revised (ADI-R) algorithm items. It has 40 yes and no questions centered around core features of ASD, and can be complete in 10-15 minutes. The SCQ shows high discriminative validity between ASD and non ASD populations, similar to the much lengthier ADI-R. ROC analyses established a cutoff score of 15 on the SCQ to differentiate between ASDs and other diagnoses. At this cutoff score, sensitivity was .85 and specificity was .75. The alpha index of internal consistency was uniform across diagnostic groups, ranging from .84 to .93. A cut off score of ≥15 will be used to corroborate a clinical diagnosis and used for inclusion. The SCQ requires 10 minutes to complete and written on 4<sup>th</sup> grade reading level.

Clinical Global Impression-Severity (CGI-S)<sup>172</sup>

This 7-point scale ranges from 1 (*Normal*) through 4 (*Moderate*) to 7 (*Extreme*). Although sleep problems will be given particular weight, independent evaluators will consider all aspects of the child's condition to assign the CGI-S score. A score of  $\geq$  4 (Moderate) is required for entry.

| Table 1. Schedule of Measures | | Baseline | <u>Wk</u> 5 | <u>Wk</u> 10 | <u>Wk</u> 16 |
|---|---|---|---|---|---|
| Parent Completed Measures | | | | | |
| Demographics, Medical & Developmental History | Χ | | | | |
| Modified Checklist for Autism in Toddlers or Social Communication<br>Questionnaire | Х | | | | |
| Composite Sleep Index (CSI) | Χ | X | Χ | Χ | X |
| Aberrant Behavior Checklist (ABC) | | Χ | Х | Χ | |
| Parent Stress Index (PSI) | | X | X | X | |
| Parenting Sense of Competence Scale (PSOC) | | Χ | Χ | Χ | |
| Parent Health Questionnaire (PHQ) | | Χ | X | Χ | |
| Pittsburgh Sleep Quality Index (PSQI) | | Χ | X | Χ | |
| Clinician Ratings | | | | | |
| Clinical Global Impressions - Severity | | Χ | X | X | |
| Clinical Global Impressions –Improvement (CGI-I) | | Χ | X | Χ | Χ |
| Safety Review | Χ | Χ | Χ | Χ | X |
| Therapist Measures | | | | | |
| Treatment Fidelity Checklists Completed at each session | | | | | |

#### Outcome Measures Sleep Measure

Composite Sleep Index (CSI) from the MSPSQ<sup>97,144,173</sup>

The CSI is a 6-item parent-report measure where items are rated 0 to 2 (range 0 to 12) with higher scores reflecting greater sleep problems. Thus, *change in an item score of 1 or 2 points reflects a clinically relevant change*. For example, for the question on frequency of night wakings, a reduction from 2 to 1 point would reflect improvement in night wakings from every night to one-two nights per week; a reduction to 0 would reflect an improvement to once a month or less. The reliability and validity of the CSI has been established as a nested scale within the MSPSQ. <sup>174</sup> Thus, we will use the full MSPSQ. Wiggs and Stores <sup>175</sup> reported the test-retest reliabilities for a 2 week period to be .83 to 1.0. In a larger study of 345 individuals with intellectual disability, Maas et al <sup>176</sup> found the internal consistency of the items of the MSPSQ to be good (Cronbach's  $\alpha$  = .80). Maas et al <sup>176</sup> also evaluated the convergent validity of the MSPSQ with a similar measure, the Sleep Disturbance Scale for Children (SDSC) and found a correlation (r = .79, p<.001) showing adequate validity. The MSPSQ has been reported to be acceptable to parents. <sup>175</sup> This measure can be completed within 5-10

minutes and is at a 5<sup>th</sup> grade reading level.

#### **Child Behavior Measures**

Improvement scale of the Clinical Global Impression (CGI-I)<sup>172</sup>

This is a clinician-rated, 7-point scale designed to measure overall improvement from baseline. Scores range from 1 (Very Much Improved) to 4 (Unchanged) to 7 (Very Much Worse). An independent evaluator (IE) **blinded** to group assignment will use all available information to judge treatment response. By convention, CGI-I ratings of Much Improved (score of 2) or Very Much Improved (score of 1) are used to classify subjects as positive responders. All other scores classify subjects as negative responders. An essential contributor to the CGI-I is the content of the semi-structured Parent Target Problem interview. <sup>31</sup> At baseline, the IE asks the parent to nominate the child's two most important problems. Based on the study entry criteria, we expect that one problem will be sleep related. The parent will also be asked to identify a second problem. Through brief discussion, the frequency (for episodic behaviors such as night wakings) or constancy (hyperactivity) reflecting more enduring patterns, intensity and impact of the behavior on the family are established. Responses from this systematic inquiry are documented in a brief narrative. The narrative will be reviewed and revised at Weeks 5, 10 and 16. This method has been shown to be reliable and valid in a previous parent training study<sup>31,177</sup> and currently being used in our RCT on parent training for feeding problems.

Aberrant Behavior Checklist. 178,179

This is a reliable and valid 58-item parent-report questionnaire with five subscales: Irritability (agitation, aggression and self-injurious behaviors), Social Withdrawal, Stereotyped Behaviors, Hyperactivity, and Inappropriate Speech. The ABC has shown adequate sensitivity to change in several pharmacological and behavioral treatment studies. The revised ABC manual science 35 scientific papers that support the convergent validity of the ABC, and its concurrent validity with several established instruments regularly used in intellectually and developmentally disabled populations. Each item is rated on a Likert scale from 0 (not a problem) to 3 (severe in degree). For the current study, we are primarily interested in change of the Irritability and Hyperactivity subscales as a proxy for sleep-related impairment (i.e., daytime behaviors secondary to sleep disturbances). Requiring an 8th grade reading level, this measure requires 15-20 minutes to complete.

#### **Quality of Life Measures**

Parenting Stress Index-Short Form (PSI)<sup>185</sup>

This is a 36-item parent-completed questionnaire for children 12 years of age and younger and has three scales: 1) Parental Distress; 2) Difficult Child Characteristics; and, 3) Dysfunctional Parent-Child Interaction. This measure was developed from the Parenting Stress Index Full Form using factor analysis, and has been used to assess parental stress and parent-child relationships in children with autism and intellectual disabilities. <sup>185-189</sup> The PSI has good test-retest reliability with an average score of .76 (min= .68, max= .85), and internal consistency (Cronbach's alpha average of .85, min= .8, max=.91). A total score of 88 (85th percentile) and above is considered in the clinically significant range for parental stress. The PSI has good convergent and concurrent validity across clinical and nonclinical samples, and diverse populations. We confirmed the factor structure in a recent study. <sup>190</sup> We have used this for several other trials and it has been shown to be sensitive to change in parent training studies. <sup>191</sup> This measure may be completed within 10-20 minutes and written at a 3rd grade reading level.

Parent Health Questionnaire-4 (PHQ-4)<sup>192</sup>

This brief self-report is designed to assess parental mental health. It has been shown to be an effective screen for anxiety and depression disorders. Requiring 5 minutes to completed and written at 5<sup>th</sup> grade reading level. The Parenting Sense of Competence scale (PSOC)<sup>193</sup>

This 17-item scale was developed to assess parental self-efficacy. Each item is answered on a 6-point scale ranging from strongly disagree to strongly agree. The measure has high internal consistency and solid test-retest reliability. The Satisfaction subscale measures parental motivation and frustration (e.g., "Even though being a parent could be rewarding, I am frustrated now while my child is at his/her present age"). The Efficacy subscale measures perceived self-efficacy to change the child's behavior (e.g., "I meet my own personal expectations for expertise in caring for my child"). The PSOC also yields a Total Competence score, with

higher scores reflecting higher competence. In a community sample of mothers, <sup>194</sup> subscale total scores of Satisfaction (22.72) and Efficacy (22.03) were reported. We have used this measure in another study of parent training and it has been shown to be sensitive to change. <sup>195</sup> This measure is written at an 8<sup>th</sup> grade reading level and requires approximately 15 minutes to complete.

#### Pittsburgh Sleep Quality Index (PSQI)<sup>196</sup>

This 19-item, self-rated questionnaire will be completed by parents. It is used in adult sleep medicine research as a reliable measure of sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime functioning. Overall, it has a reliability coefficient (Cronbach's alpha) of 0.83, indicating a high degree of internal consistency. For the subgroup that was tested at two time points, the correlation coefficient for global PSQI scores was 0.85 (p<0.001). Distribution of global PSQI scores differed between groups. A cutoff score of 5 correctly identified 88.5% of all patients and controls (kappa=0.75, p<0.001). This represents a sensitivity of 89.6% and a specificity of 86.5%. PSQI estimates of sleep variables were compared to polysomnographic findings. T-tests showed no differences between PSQI sleep latency estimates and those found using polysomnography, but estimates of usual sleep duration and efficiency were greater than those obtained through polysomnography. The reading level for this widely used measure is written at the 3rd-4<sup>th</sup> grade reading level and requires around 10 minutes.

#### **Clinician Measures**

#### Treatment Fidelity Checklist

These checklists include the therapist integrity goals, parent objectives and level of adherence for each SPT and SPE session. Therapists rate themselves on 5-7 session-specific goals on a scale of 0 to 2 as follows: (0 = Goal was not achieved; 1 = Goal was partially achieved; 2 = Goal was fully achieved). Therapists are asked to comment on items rated 0. Parent objectives and adherence are scored on a similar scale. The score for each session = sum of scores for all items in that session divided by the total possible score X 100. An example of a treatment fidelity checklist is in Intervention section. These treatment fidelity checklists have been modeled after four other previously NIH-funded projects.  $^{31,97,148,191}$ 

# Safety/Adverse Event Review Form

Starting at the screen visit, the masked Independent Evaluator (IE) will ask about recent health complaints, use of medical services and concomitant medications. The Safety/Adverse Event Review Form also asks about the child's sleep, appetite and bowel habits. Screen data will be documented so that new adverse events can be elicited and recorded using the same Safety/Adverse Event Review Form. Reports of new adverse events or worsening of previously reported events will be rated mild (present, but not a problem), moderate (present, posing a problem or intervention required to prevent a problem) or severe (present, posing a problem and needed intervention). Hospitalization will be documented as a serious adverse event. A "yes" answer to any of these queries will prompt further questions to determine duration and severity. The onset, offset and severity of adverse events will be documented whether presumed to be related to the study treatment or not (see Human Subjects section).

# **Description of Interventions**

#### **Behavioral Parent Training for Sleep Disturbances (SPT)**

SPT is an expanded version of the single sleep session that the PI (C. Johnson) developed for the RUPP Autism Network Parent Training (PT) program (U10MH66764] and the recently completed Research Units on Behavioral Intervention PT program [RUBI, R01MH1081148MH; Johnson, PI). 31,197,198 SPT was developed and evaluated for feasibility and initial test of efficacy (R34MH08288: Johnson, PI). 7 The five SPT sessions (each 60-90 minutes in duration) are individually delivered over 10-weeks (see Table 2). In addition to the five sessions, there are three home visits conducted via Express Care Online (HIPAA compliant video-chat). After Session A, session order may be adjusted to address child-specific problems. For example, if night wakings is the highest priority, Session C may be offered before Session B to introduce the use of extinction or scheduled wakings. Spreading the sessions over 10 weeks allows for scheduling flexibility and opportunities to present child-specific optional materials (outlined in Table 2). All parents/caregivers who are involved with the child's bedtime and sleep will be encouraged to participate. Hopefully, telehealth delivery will facilitate fuller

inclusion of caregivers. Each session employs direct instruction, modeling, and role-playing to promote parental skill acquisition. The SPT manual includes a therapist script and parent activity sheets for each session. Video vignettes have been developed for each session that model specific techniques and show a parent incorrectly applying the technique for different bedtime problems. For example, vignettes show a parent reacting to a child's tantrum at bedtime and a parent responding to a child calling out in the middle of the night. By showing ineffective parent management strategies, the video vignettes supplement direct instruction. In discussion, the parent is encouraged to identify the error in the vignette and to consider alternative responses. Thus, the video vignettes serve as a check on the parents' acquisition of concepts and techniques and permit the therapist to clarify uncertainties. Parents are given homework assignments to practice new skills learned in each session along with data collection assignments. The materials from one of the SPT session are provided in the Intervention section.

#### Rationale for SPT

Parent training based on the principles of applied behavior analysis is an empirically supported intervention for

| Table 2. SPT Session Out | |
|---|---|
| Sessions | Topics Addressed |
| A. Importance of Sleep &<br>Basic Behavioral<br>Principles | <ul> <li>Introduce overall goals.</li> <li>Introduce importance of sleep and the need to improve quality of sleep in children with ASD.</li> <li>Introduce antecedent, behavior, and consequence model.</li> <li>Introduce the concept of the functions of behavior.</li> <li>Introduce general sleep hygiene guidelines.</li> <li>View bedroom / sleeping environment</li> </ul> |
| B. Addressing<br>Prevention Techniques &<br>Bedtime Routines | <ul> <li>Discuss preventive techniques .specific to children with ASD.</li> <li>Develop daily schedule as well as bedtime schedule / routine.</li> <li>Develop visual schedule that supports daily/bedtime routine.</li> <li>Review how to develop social stories, when appropriate.</li> </ul> |
| VSEE Evening Session | Parent coaching at bedtime |
| C. Addressing the Use of<br>Extinction & Procedures<br>for Bedtime Struggles,<br>Night Wakings and Early<br>Morning Wakings | <ul> <li>Introduce concept of extinction / planned ignoring to decrease behaviors.</li> <li>Introduce use of different extinction techniques to specifically address sleep problems (bedtime struggles, night wakings, early morning wakings).</li> <li>Introduce concept of reinforcers and teach contingent implementation of reinforcement.</li> <li>Decide upon reinforcement, extinction, &amp; scheduled awakening procedures.</li> </ul> |
| VSEE Evening Session | Parent coaching at bedtime |
| D. Addressing Delayed<br>Sleep Onset & Sleep<br>Association Procedures | <ul> <li>Introduce the concept of stimulus control and its relationship to sleep behaviors.</li> <li>Introduce faded bedtime routines as well as review bedtime routine.</li> <li>Introduce teaching new sleep associations.</li> <li>Develop specific procedures for teaching new sleep associations.</li> </ul> |
| VSEE Evening Session | Parent coaching at bedtime |
| E. Booster &<br>Maintenance Session | <ul> <li>Revise &amp; "tweak" procedures / techniques based on review of sleep diary data and parent report of progress.</li> <li>Discuss strategies for maintenance of behavior change.</li> <li>Generate ideas of what to do if changes do not / have not maintained.</li> </ul> |
| OPTIONAL MATERIALS<br>Address Noncompliance | Introduce concept of compliance / noncompliance Review steps for compliance training Review procedures for increasing compliance around bedtime and nighttime |
| Address Nighttime Fears | <ul> <li>Review why children may have fears at nighttime</li> <li>Discuss with parent's their child's fears</li> <li>Develop plan to reassure child, teach the child "brave skills"</li> <li>Teach parents to implement systematic exposure for severe/specific fears</li> </ul> |


young children with ASD and disruptive behavior.<sup>31</sup> For sleep problems, parent training was also chosen for pragmatic reasons: a parent/caregiver is available at bedtime when sleep disturbances occur; and parents (and other family members) may be adversely affected by the child's sleep disturbance. The decision to have all participants complete the five-session SPT program, regardless of primary sleep complaint is based on the observation that children with ASD often have more than one sleep problem and sleep problems can change over time in this population.<sup>97</sup> Thus, SPT provides a comprehensive intervention that teaches parents the basic concepts and practical skills to address an array of sleep problems. One-on-one delivery of SPT permits flexibility for child-specific problems within the program.

#### Rationale and Modifications of SPT for Telehealth Delivery.

Telehealth delivery of SPT is expected to not only be more feasible in that it will allow families who live a distance from tertiary, specialized autism centers to participate, but is more optimal in that materials from the sessions may be delivered at a time more convenient for them; even soon before bedtime so content is fresh for parents. This will also allow us to complete more parent-child coaching in this manner of delivery. Overall, ecological validity of the intervention will be enhanced by delivering SPT via telehealth platform. Modifications to be made to allow for telehealth delivery are minimal. Session activity sheets the parents will need will be pushed out by REDCap ahead of time. Hard copies will also be mailed if families prefer. The video vignettes used in each session will be viewed via the split screen of Express Care Online. We can also provide the families with a DVD of the videos if they wish. Materials that might have been developed in session for the family to use at home (for example, a visual schedule) will be overnight mailed to the family as well as pushed out to them by REDCap link.

#### **Sleep Parent Education (SPE)**

SPE consists of five 60-90 minute sessions, delivered individually over 10 weeks. As with SPT, we expect one parent to attend all sessions, but another parent or caregiver is invited to attend SPE. As shown in Table 3, SPE provides useful information to families of young children with ASD and sleep problems. Session A is designed to develop rapport. The sleep hygiene session (Session B) has been modeled from the RUBI manual. The other

| Table 3. Sleep Hygiene a | and Parent Education (SPE) Outline |
|---|---|
| Sessions | Goals & Topics Addressed |
| A. ASD Diagnosis | <ul> <li>Discuss diagnosis &amp; family's adjustment</li> </ul> |
| _ | <ul> <li>Prevalence of ASD in the population and etiology</li> </ul> |
| | Review service delivery models |
| | <ul> <li>Review sleep diary to be completed for next session</li> </ul> |
| B. Sleep Hygiene | <ul> <li>Introduce types of sleep disturbances observed in ASD</li> </ul> |
| | <ul> <li>Review CSI and Sleep Diary with parent(s)</li> </ul> |
| | <ul> <li>Develop plan to address identified bedtime / sleep problems</li> </ul> |
| | <ul> <li>Develop data collection to monitor progress</li> </ul> |
| C. Understanding & | <ul> <li>What do IQ tests measure &amp; understanding the scores</li> </ul> |
| Interpreting Clinical | <ul> <li>Speech, language and communication measures</li> </ul> |
| Evaluations | Fine motor measures |
| | <ul> <li>Review selected behavioral ratings</li> </ul> |
| D. Advocacy and | <ul> <li>Provide information about national &amp; local support services</li> </ul> |
| Support Services | Parent to parent contact |
| | <ul> <li>Advocacy services and how to use them</li> </ul> |
| E. Treatments & | <ul> <li>Information on evidence-based / best practices</li> </ul> |
| Treatment Planning | <ul> <li>Information on other alternative treatments &amp; use of<br/>supplements</li> </ul> |
| | Review of current services for child |
| | Discuss progress and current concerns |
| | Discuss other treatment options available for children with ASD |


sessions include a systematic presentation on several relevant topics (see Table 3). An example of a SPE session is provided in the Intervention section. This control condition is intended to parallel what would be offered in typical care, but by telehealth, where a parent might be educated about ASD as well as attend an outpatient appointment at a sleep clinic.

#### Rationale for SPE as the control condition

SPE is a structured program intended to mimic competent *treatment as usual*. Thus, SPE is an accepted treatment and serves as an active comparator that controls for time and attention. We have conducted two previous randomized trials using parent education as the control condition. In both studies, attrition was low and satisfaction was high.<sup>31,97</sup>

Rationale and Modifications of SPE for Telehealth Delivery. Given our success with using SPE as an active comparator in previous studies, we are optimistic about using this control for the current study. As with SPT, minimal modifications will need to be made to deliver SPE individually via telehealth platform. All materials parents will need for SPE will be pushed out via REDCap, with the option of a hard copy mailed to them as well. In fact, telehealth delivery of SPE is more interactive than many internet-based programs that parents use to seek knowledge about ASD (e.g. Autism Speaks, Autism Navigator, Organization for Autism Research). Parents in SPE will receive the benefits of a therapist to respond to their specific questions and as aforementioned, parents in previous trials have been extremely satisfied with SPE. 31,97

# **Quality Control**

#### Assessments

Measures to be used for this study have all been used in prior studies by Dr. Johnson. At a start up meeting, the research team will review all measures. Dr. Johnson will review with independent evaluators (IEs) on the elicitation and documentation of the Parent Target Problems specifically around and to use all available information to rate the CGI-S and CGI-I, and to conduct the Safety/Adverse Event Review.

### Therapist Selection, Training & Fidelity Monitoring

Doctoral or masters level practitioners with behavioral intervention experience in children with ASD will provide study treatments. Dr. Johnson, who has extensive therapist training experience, will train study therapist(s). Therapists will read through the treatment manual and observe sessions (or videos) by an experienced clinician delivering SPT and SPE. Similar to our other studies, therapists will be trained to 80% reliability for each session of both manuals with a non-study subject prior to treating randomized study subjects. The reliability will be confirmed by review of audio recordings by Dr. Johnson. After each SPT or SPE session, therapists will rate their own fidelity on a set of session-specific goals using a 0-2 scale (0=item not covered, 1=partially covered, 2=fully covered). All sessions in the randomized trial will be audio recorded and a 10% sample of randomly selected recordings will be scored to monitor therapist fidelity throughout the study. If therapist fidelity falls below criterion, a remedial plan will be implemented. Another element of treatment integrity is parental adherence (compliance and engagement). Therapists will rate parental adherence to SPT or SPE on a similar 0 to 2 scale. Parental adherence that falls below 70% in two successive sessions will be directly discussed with the parent. A session treatment fidelity form example may be found in the Intervention section along with session materials.

# **Data Management and Analyses**

#### **Data Management**

Data will be collected directly via the web-based data entry site, developed through REDCap. <sup>171</sup> REDCap is a secure, web-based application for building and managing online surveys and databases. The REDCap software, training videos and basic end-user support are provided to all Cleveland Clinic investigators without charge. The system is managed by the Cleveland Clinic Center for Clinical Research and Learner Research Institute Research Computing Services. REDCap resides on servers within the Learner Research Institute. This centrally-located data center features redundant, high availability infrastructure components, including over 100TB of XIOTech SAN and SATA storage capacity, IBM Tivoli tape libraries for backup, HP servers, VMWare Virtual Infrastructure Clusters and a system-wide Liebert 130KVA Uninterrupted Power Supply. Data are backed up hourly at 3 separate, secure locations.

Page **14** of **27** 

Data management analyst (TBN) under the direction of biostatistician (Sarah Worley) will develop the online data collection forms through REDCap. The data entry forms will be designed with as few open-ended text fields, and as many user-friendly drop-down answer boxes or check boxes as possible, with little opportunity for responses to be provided with implausible values. Clinic data will be entered by the study coordinators; the entry forms will be developed with built-in range checks and automatically-calculated fields to reduce the possibilities of data entry errors. Branching logic will be extensively used so questions/fields do not need to appear when they are illogical. The database will be pilot-tested after development, with feedback from the coordinator on ease of use. A separate randomization assignment data set will exist with a common identifier to allow for linkage with the study database for final analyses. This randomization data set will be maintained on a secure server and only accessible by the data management team. During enrollment, the data manager will regularly check for data inconsistencies, omissions, and errors, confirming with the coordinator when outliers and unusual values are observed. The data manager will randomly select 10% of data on a quarterly basis to be checked for data entry quality; discrepancies will trigger review of data collection and entry procedures as appropriate. The data management team will attend all study meetings to ensure constant communication about data issues that may arise throughout the study.

#### Sample Size and Power Calculation for Primary Hypotheses.

We base our power analysis on the primary aim/analysis comparing efficacy of SPT for sleep disturbance in children with ASD compared to SPE, with the CSI score as the primary outcome. Specifically, we aim to achieve 90% power to detect a meaningful difference in change in CSI scores between baseline and 10 weeks between the SPT and SPE groups ( $\alpha = 0.05$ ). We assume we will have roughly 40 participants per group (80 total) after allowing for an attrition rate of about 10% in each group as has been average from our previous clinical trials. A 2-point difference in the CSI score (CSI description below) is clinically relevant. Based on our preliminary study (Figure 1), we observed a SD = 2.5 for the difference between baseline and 8-week CSI scores in the treatment group and a SD = 2.3 for the difference in the control group. The SD's for the 4-week difference were also equal to 2.3 in both groups; thus a conservative SD estimate of 2.5 for the difference between baseline and 10 weeks was used. For the parameters listed above and a total final sample size of 80, we will have 90% power to detect a difference in 10-week CSI change of 1.7 points or greater. Given the constant SD's observed over time, this power analysis is reasonable for 5-week comparisons as well. For hypothesis 2, specifically focusing on the CGI-I, we predict somewhere between 25%-40% positive response in the SPE group. With 45 per group (CGI-I drop-outs will be classified as negative responders by default), we will have 90% power ( $\alpha$ =0.05) to detect a 32% or greater difference in positive response rate (57%-72%, respectively).

#### **Statistical Analysis**

Statistical analyses will be conducted by Sarah Worley in collaboration with the study team. We will begin with descriptive statistics for baseline data across treatment groups. Study coordinator and data manager will inspect data for errors, inconsistencies, and incomplete information across time points (as a follow-up to the regular data management procedures that will occur throughout the study, described above). This will include examination of frequency tables and scatter plots. Data anomalies and outliers will be examined and corrected if necessary. These preliminary analyses will include descriptive statistics in each treatment group for all outcome variables, plots of longitudinal data over time, and examination of distributions within groups at important nodal points (e.g., Baseline, Week 5, 10 and 16). For the **primary analysis**, we will use a linear mixed model, which will make use of the repeated measurement of the CSI. Specifically, we will model change in CSI relative to baseline at weeks 5 and 10 (and week 16), with primary fixed effects of baseline CSI, treatment (SPT or SPE), time, and the interaction between time and treatment. No systematic trend with time will be initially assumed to allow for potential nonlinear trends; if linear changes are observed (and confirmed via statistical testing), we will model time as a continuous variable. With at most three repeated measurements, model selection of the covariance structure is minimized; we will model directly the variance of the outcome at each time point as well as the correlation between the three visits (i.e., unstructured covariance). We will examine whether the covariance needs to be modeled separately between the two treatment groups, as well as whether


we can use a more parsimonious covariance model to maximize statistical power. Common model selection criteria will be used for this examination. Appropriate assumptions and model conditions will be verified prior to analysis. Tabled data will be presented as differences in means across time with 95% confidence intervals. The Kenward-Roger approximation for the denominator degrees of freedom will be utilized to ensure valid inference of the fixed effects. A similar approach will be used for the key continuous secondary outcome (Total Sleep Time on actigraph) and other secondary measures such as the ABC- Irritability subscale, PSI scales, Parental Competence measure, etc. The **key secondary analysis** will use the chi-square test to compare the rate of positive response on the CGI-I in SPT versus SPE. Chi-square tests will also be used to compare the rates of adverse events across treatment groups.

Efficacy analyses will follow the *intention-to-treat* convention (including all randomized subjects). For modeling and hypothesis testing, the proposed likelihood-based approach regards missing data as missing at random (MAR; i.e., missing data are independent of unobserved data). Although there is no proven method for verifying the MAR assumption, the likelihood-based solutions are robust to violations of ignorable missing data (i.e., situations where the MAR assumption is not met). Prior to analyses for efficacy, we will examine the degree of randomness in missing data by comparing the frequency, reasons, pattern and time to dropout and missing values across treatment groups. If substantial differences in *missingness* occur across SPT and SPE that cannot be adequately explained by observed variables, secondary sensitivity analyses employing the methods described by Carpenter and Kenward<sup>202</sup> will be employed. These techniques will be considered cautiously in our analyses as they require certain assumptions that cannot be evaluated from the data under analysis. All analyses will be conducted using SAS v9.4 for Windows (Cary, NC, USA).

Given the planned sample size, we will not have sufficient statistical power to detect effect modifiers (i.e., compare the efficacy of the intervention among subgroups). However, we do plan to examine and compare the efficacy of the intervention between subgroups via statistical interactions in the above models. Variables of interest include age, IQ, and gender. These estimates, if we observe possible differential effects, will serve as the basis for future, larger studies that target the comprehensive study by subgroups.

The above general analysis plan holds for the majority of our aims/hypotheses. We discuss specifics analysis considerations below for each aim/hypothesis as appropriate.

#### **Primary Aim**

To evaluate the efficacy of telehealth delivery of SPT for sleep disturbance in children with ASD compared to telehealth delivery of SPE.

<u>Hypothesis 1</u>: After 10 weeks of treatment, children whose parents receive SPT will show greater reduction on the CSI from the MSPSQ compared to those whose parents receive SPE. *Our modeling approach above describes how we will test this hypothesis, with change in CSI relative to baseline as our outcome to be modeled over the span of the study via linear mixed models (5 and 10 weeks).* 

<u>Hypothesis 2</u>: After 10 weeks of treatment, children in the SPT group will show significantly higher rates of positive response than children in the SPE group on the Improvement scale of the Clinical Global Impression (CGI-I) rated by an independent evaluator masked to group assignment. *The proportion of positive response (Much Improved or Very Much Improved) in SPT vs SPE will be tested using a Chi Square test.* 

<u>Hypothesis 3</u>: After 10 weeks of treatment, children whose parents receive SPT will show significantly lower rates of disruptive behaviors on the parent-rated ABC-Irritability subscale compared to children whose parents receive SPE. *To test this hypothesis, we will use the same linear mixed model approach described for the CSI*. The other ABC subscales will be examined in exploratory analyses.

Hypothesis 4: As noted above, all subjects will be asked to return at Week 16 to evaluate the post-treatment effects of SPT and SPE. Parents will rate the CSI. The same treatment blinded IE will rate the CGI-I at post-treatment follow up. We will essentially add the 16-week CSI measure to the modeling framework described above to further characterize CSI trends over a longer period of time, and to compare these trends between the two groups. This modeling approach (in particular modeling the time point directly (i.e., not assuming a linear trend from baseline) will allow us to directly test for differences at 16 weeks. We will also compare the rate of

positive response on the CGI-I in the SPT versus SPE. Subjects who drop out before or after Week 10 will be classified as negative responders by default.

# **Secondary Aim**

To evaluate the impact of SPT on parental quality of life (parental stress, sense of competence, mental health and sleep) compared to SPE.

<u>Hypothesis 1 and 2</u>: After 10 Weeks of treatment, parents in SPT will report lower levels of stress and higher levels of competency and overall health as measured by the PSI (stress), PSOC (competence), PHQ (mental health) and better PSQI (sleep) than parents in SPE. To test these hypotheses, we will use the same linear mixed model approach described for the CSI. Exploratory analyses will test whether parental quality of life shows greater change from baseline to week 16 on the PSI, PSOC, PSQ, and PSQI compared to SPE.

# **Timetable of Projected Activities**

A total of 90 children will be recruited. In the second half of Year 01, each site will screen 17-18 subjects with the goal of randomizing 15 subjects. In Years 2 and 3, we aim intend to randomize 30 subjects per year. In the first half of Year 04, we will

| Table 4. Timetable | Month<br>0-6 | Month 6-<br>12 | Year 02 | Year 03 | Year 04 |
|---|---|---|---|---|---|
| IRB approval finalized | Х | | | | |
| Set Up Entry Programs | Х | | | | |
| Train Therapists | Х | | | I | |
| Recruitment & Enrollment | | X | X | X | X |
| Conduct Interventions | | X | X | X | X |
| Follow-Up Assessments | | X | X | X | X |
| Data Analysis | | | | | X |
| Manuscript Preparation | | 0 | Į. | | X |
| Dissemination | | | | T) | X |

screen 17-18 subjects to meet goal of randomizing the final 15 participants (see Table 4).

#### References

- 1. Elsabbagh M, Divan G, Koh YJ, et al. Global prevalence of autism and other pervasive developmental disorders. *Autism Research*. 2012;5(3):160-179.
- 2. Christensen DL, Baio J, Van Naarden Braun K, et al. Prevalence and characteristics of autism spectrum disorder among children aged 8 years—autism and developmental disabilities monitoring network, 11 sites, United States, 2012. *MMWR Surveillance Summaries*. 2016;65(3):1-23.
- 3. Brereton AV, Tonge BJ, Einfeld SL. Psychopathology in children and adolescents with autism compared to young people with intellectual disability. *Journal of Autism and Developmental Disorders*. 2006;36(7):863-870.
- 4. Hartley S, Sikora D, McCoy R. Prevalence and risk factors of maladaptive behaviour in young children with autistic disorder. *Journal of Intellectual Disability Research*. 2008;52(10):819-829.
- 5. Lecavalier L. Behavioral and emotional problems in young people with pervasive developmental disorders: Relative prevalence, effects of subject characteristics, and empirical classification. *Journal of Autism and Developmental Disorders*. 2006;36(8):1101-1114.
- 6. Rosenberg RE, Kaufmann WE, Law JK, Law PA. Parent report of community psychiatric comorbid diagnoses in autism spectrum disorders. *Autism research and treatment*. 2011;2011.
- 7. Simonoff E, Pickles A, Charman T, Chandler S, Loucas T, Baird G. Psychiatric disorders in children with autism spectrum disorders: Prevalence, comorbidity, and associated factors in a population-derived sample. *Journal of the American Academy of Child & Adolescent Psychiatry*. 2008;47(8):921-929.
- 8. Hallett V, Lecavalier L, Sukhodolsky D, et al. Exploring the Manifestations of Anxiety in Children with Autism Spectrum Disorders. *Journal of Autism and Developmental Disorders*. 2013;43(10):2341-2352.
- 9. Honomichl RD, Goodlin-Jones B, Burnham MM, Gaylor E, Anders T. Sleep patterns of children with pervasive developmental disorders. *Journal of Autism and Developmental Disorders*. 2002;32(6):553-561.
- 10. Johnson CR. Sleep problems in children with mental retardation and autism. *Child and Adolescent Psychiatric Clinics of North America*. 1996;5(3):673–683.
- 11. Johnson CR, Turner KS, Foldes EL, Malow BA, Wiggs L. Comparison of sleep questionnaires in the assessment of sleep disturbances in children with autism spectrum disorders. *Sleep Medicine*. 2012;13(7):795-801.
- Wiggs L, Stores G. Sleep patterns and sleep disorders in children with autistic spectrum disorders: insights using parent report and actigraphy. *Developmental Medicine & Child Neurology*. 2004;46(6):372-380.
- 13. Coury D. Medical treatment of autism spectrum disorders. *Current opinion in neurology*. 2010;23(2):131-136.
- 14. Knapp M, Mandell D, Buescher A, Cidav A. Autism: Economic impact and implications. *Autism Summit, Investing in our Future.* 2012.
- 15. Rogers SJ, Vismara LA. Evidence-based comprehensive treatments for early autism. *Journal of Clinical Child & Adolescent Psychology.* 2008;37(1):8-38.
- 16. Sallows GO, Graupner TD. Intensive behavioral treatment for children with autism: Four-year outcome and predictors. *American Journal of Mental Retardation*. 2005;110(6):417-438.
- 17. Smith T, Scahill L, Dawson G, et al. Designing Research Studies on Psychosocial Interventions in Autism. *Journal of Autism and Developmental Disorders*. 2007;37(2):354-366.
- 18. Prizant BM, Wetherby AM, Rubin E, Laurent AC, Rydell PJ. *The SCERTS [TM] Model: A Comprehensive Educational Approach for Children with Autism Spectrum Disorders*. ERIC; 2005.


- 19. Council NR. Educating children with autism. Committee on Educational Interventions for Children with Autism. In: Lord C, McGee JP, eds. *Division of Behavioral and Social Sciences and Education*. Washington, DC:: National Academy Press; 2001.
- 20. Matson JL, Dempsey T. Autism spectrum disorders: Pharmacotherapy for challenging behaviors. *Journal of Developmental and Physical Disabilities*. 2008;20(2):175-191.
- 21. Scahill L, Martin A. Psychopharmacology. In: Volkmar F, Klin A, Paul R, eds. *Handbook of Autism and Pervasive Developmental Disorders* 3rd ed. New York: Wiley; 2005:1102-1117.
- 22. Croen LA, Grether JK, Hoogstrate J, Selvin S. The changing prevalence of autism in California. *Journal of Autism and Developmental Disorders*. 2002;32:207-215.
- 23. Gerhardt PF, Lainer I. Addressing the needs of adolescents and adults with autism: a crisis on the horizon. *Journal of Contemporary Psychotherapy*. 2011;41(1):37-45.
- 24. Jensen VK, Sinclair LV. Treatment of autism in young children: behavioral intervention and applied behavior analysis. *Infants & Young Children*. 2002;14(4):42-52.
- 25. Stahmer A. The Basic Structure of Community Early Intervention Programs for Children with Autism: Provider Descriptions. *Journal of Autism and Developmental Disorders*. 2007;37(7):1344-1354.
- 26. Committee IAC. IACC strategic plan for autism spectrum disorder research. *Washington (DC): US Department of Health and Human Services.* 2011.
- 27. Organization WH. *Atlas: Global resources for persons with intellectual disabilities 2007.* World Health Organization; 2007.
- 28. Brookman-Frazee L, Drahota A, Stadnick N, Palinkas LA. Therapist perspectives on community mental health services for children with autism spectrum disorders. *Administration and Policy in Mental Health and Mental Health Services Research*. 2012;39(5):365-373.
- 29. Meltzer LJ, Phillips C, Mindell JA. Clinical psychology training in sleep and sleep disorders. *Journal of Clinical Psychology*. 2009;65(3):305-318.
- 30. Wacker DP, Lee JF, Dalmau YCP, et al. Conducting functional analyses of problem behavior via telehealth. *Journal of Applied Behavior Analysis*. 2013;46(1):31-46.
- 31. Bearss K, Johnson, C.R., Smith, T. . Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: A randomized clinical trial. *Journal of the American Medical Association*. 2015;313(15):1524-1533.
- 32. Garstang J, Wallis M. Randomized controlled trial of melatonin for children with autistic spectrum disorders and sleep problems. *Child: Care, Health, and Development.* 2006;32(5):585-589.
- 33. Iglowstein I, Jenni OG, Molinari L, Largo RH. Sleep duration from infancy to adolescence: Reference values and generational trends. *Pediatrics*. 2003;111(2):302-307.
- 34. Moore M, Allison D, Rosen CL. A review of pediatric nonrespiratory sleep disorders. *Chest.* 2006;130(4):1252-1262.
- 35. Meltzer LJ, Mindell JA. Sleep and sleep disorders in children and adolescents. *Psychiatric Clinics of North America*. 2006;29(4):1059-1076.
- 36. Stores GE, Wiggs LE. *Sleep disturbance in children and adolescents with disorders of development: Its significance and management.* Cambridge University Press; 2001.
- 37. Stores G. Sleep-wake function in children with neurodevelopmental and psychiatric disorders. *Seminars in Pediatric Neurology*. 2001;8(4):188-197.
- 38. Dahl RE. The impact of inadequate sleep on children's daytime cognitive function. *Seminars in Pediatric Neurology*. 1996;3(1):44-50.
- 39. Graven S. Sleep and brain development. *Clinics in Perinatology*. 2006;33(3):693.
- 40. Kurth S, Ringli M, Geiger A, LeBourgeois MK, Jenni OG, Huber R. Mapping of Cortical Activity in the First Two Decades of Life: A High-Density Sleep Electroencephalogram Study. *Journal of Neuroscience*, 2010;30(40):13211-13219.
- 41. Bernier A, Carlson SM, Bordeleau S, Carrier J. Relations between physiological and cognitive regulatory systems: Infant sleep regulation and subsequent executive functioning. *Child Development*. 2010;81(6):1739-1752.

- 42. Frank MG, Issa NP, Stryker MP. Sleep enhances plasticity in the developing visual cortex. *Neuron*. 2001;30(1):275.
- 43. Goel N, Rao H, Durmer JS, Dinges DF. Neurocognitive consequences of sleep deprivation. *Semin Neurol.* 2009;29(4):320-339.
- 44. Maquet P. The Role of Sleep in Learning and Memory. *Science*. 2001;294(5544):1048-1052.
- 45. Sadeh AVI, Gruber R, Raviv A. Sleep, neurobehavioral functioning, and behavior problems in schoolage children. *Child Development*. 2002;73(2):405-417.
- 46. Stickgold R, Walker MP. Sleep and memory: the ongoing debate. *Sleep.* 2005;28(10):1225-1227.
- 47. Walker MP, Stickgold R. Sleep, memory, and plasticity *Annual review of psychology*. 2006;57(1):139-166
- 48. Leotta C, Carskadon M, Acebo C, Seifer R, Quinn B. Effects of acute sleep restriction on affective response in adolescents: Preliminary results. *Sleep Research*. 1997;26:201.
- 49. Randazzo AC, Muehlbach MJ, Schweitzer PK, Walsh JK. Cognitive function following acute sleep restriction in children ages 10-14. *Sleep: Journal of Sleep Research & Sleep Medicine*. 1998.
- 50. Steenari M-R, Vuontela V, Paavonen EJ, Carlson S, Fjällberg M, Aronen ET. Working memory and sleep in 6-to 13-year-old schoolchildren. *Journal of the American Academy of Child & Adolescent Psychiatry*. 2003;42(1):85-92.
- 51. Vriend JL, Davidson FD, Corkum PV, Rusak B, McLaughlin EN, Chambers CT. Sleep quantity and quality in relation to daytime functioning in children. *Children's Health Care*. 2012;41(3):204-222.
- 52. Sadeh A, Gruber R, Raviv A. The effects of sleep restriction and extension on school-age children: What a difference an hour makes. *Child Development*. 2003;74(2):444-455.
- 53. Fallone G, Acebo C, Arnedt JT, Seifer R, Carskadon MA. Effects of acute sleep restriction on behavior, sustained attention, and response inhibition in children. *Perceptual and Motor Skills* 2001;93(1):213-229.
- 54. Fallone G, Acebo C, Seifer R, Carskadon MA. Experimental restriction of sleep opportunity in children: effects on teacher ratings. *Sleep.* 2005;28(12):1561.
- 55. Gruber R, Grizenko N, Schwartz G, Bellingham J, Guzman R, Joober R. Performance on the continuous performance test in children with ADHD is associated with sleep efficiency. *Sleep.* 2007;30(8):1003.
- 56. Gruber R, Xi T, Frenette S, Robert M, Vannasinh P, Carrier J. Sleep disturbances in prepubertal children with attention deficit hyperactivity disorder: a home polysomnography study. *Sleep.* 2009;32(3):343.
- 57. Gruber R, Cassoff J, Frenette S, Wiebe S, Carrier J. Impact of sleep extension and restriction on children's emotional lability and impulsivity. *Pediatrics*. 2012;130(5):e1155-e1161.
- 58. Gruber R, Wiebe S, Montecalvo L, Brunetti B, Amsel R, Carrier J. Impact of sleep restriction on neurobehavioral functioning of children with attention deficit hyperactivity disorder. *Sleep*. 2011;34(3):315.
- 59. Peters JD, Biggs SN, Bauer KM, et al. The sensitivity of a PDA- based psychomotor vigilance task to sleep restriction in 10- year- old girls. *Journal of Sleep Research*. 2009;18(2):173-177.
- 60. Fredriksen K, Rhodes J, Reddy R, Way N. Sleepless in Chicago: tracking the effects of adolescent sleep loss during the middle school years. *Child Development*. 2004;75(1):84-95.
- 61. Gregory AM, Rijsdijk FV, Eley TC. A twin study of sleep difficulties in school aged children. *Child Development*. 2006;77(6):1668-1679.
- 62. Kurnatowski P, Putyński L, Łapienis M, Kowalska B. Physical and emotional disturbances in children with adenotonsillar hypertrophy. *The Journal of Laryngology & Otology*. 2008;122(09):931-935.
- 63. Carskadon MA, Harvey K, Dement WC. Sleep loss in young adolescents. *Sleep.* 1981;4(3):299-312.
- 64. Wolfson AR, Carskadon MA. Sleep schedules and daytime functioning in adolescents. *Child Development*. 1998;69(4):875-887.
- 65. Bates JE, Viken RJ, Alexander DB, Beyers J, Stockton L. Sleep and adjustment in preschool children: Sleep diary reports by mothers relate to behavior reports by teachers. *Child Development*. 2002;73(1):62-75.
- 66. Chu J, Richdale AL. Sleep quality and psychological wellbeing in mothers of children with developmental disabilities. *Research in Developmental Disabilities*. 2009;30(6):1512-1522.

- 67. Couturier JL, Speechley KN, Steele M, Norman R, Stringer B, Nicolson R. Parental perception of sleep problems in children of normal intelligence with pervasive developmental disorders: prevalence, severity, and pattern. *Journal of American Academy of Child and Adolescent Psychiatry*. 2005;44(8):815-822.
- 68. Wiggs L, Stores G. Behavioural treatment for sleep problems in children with severe intellectual disabilities and daytime challenging behaviour: Effect on mothers and fathers. *British Journal of Health Psychology*. 2001;6(3):257.
- 69. Alfano CA, Ginsburg GS, Kingery JN. Sleep-related problems among children and adolescents with anxiety disorders. *Journal of the American Academy of Child & Adolescent Psychiatry*. 2007;46(2):224-232.
- 70. Scott N, Blair PS, Emond AM, et al. Sleep patterns in children with ADHD: a population-based cohort study from birth to 11 years. *Journal of Sleep Research*. 2013;22(2):121-128.
- 71. Dahl R, Lewin D. Sleep and depression. In: G.Stores, L.Wiggs, eds. *Sleep disturbance in children and adolescents with disorders of development: Its significance and management*. New York: Cambridge University Press; 2001:161–168.
- 72. Glod CA, Teicher MH, Hartman CR, Harakal T. Increased nocturnal activity and impaired sleep maintenance in abused children. *Journal of the American Academy of Child & Adolescent Psychiatry*. 1997;36(9):1236-1243.
- 73. Gregory AM, Caspi A, Eley TC, Moffitt TE, O'Connor TG, Poulton R. Prospective longitudinal associations between persistent sleep problems in childhood and anxiety and depression disorders in adulthood. *Journal of Abnormal Child Psychology*. 2005;33(2):157-163.
- 74. Gregory AM, Rijsdijk FV, Dahl RE, McGuffin P, Eley TC. Associations between sleep problems, anxiety, and depression in twins at 8 years of age. *Pediatrics*. 2006;118(3):1124-1132.
- 75. Harvey AG. Sleep and circadian rhythms in bipolar disorder: Seeking synchrony, harmony, and regulation. *The American Journal of Psychiatry*. 2008;165(7):820-829.
- 76. El- Sheikh M, Buckhalt JA, Mark Cummings E, Keller P. Sleep disruptions and emotional insecurity are pathways of risk for children. *Journal of Child Psychology and Psychiatry*. 2007;48(1):88-96.
- 77. Smaldone A, Honig JC, Byrne MW. Does assessing sleep inadequacy across its continuum inform associations with child and family health? *Journal of Pediatric Health Care*. 2009;23(6):394-404.
- 78. Gregory AM, Van der Ende J, Willis TA, Verhulst FC. Parent-reported sleep problems during development and self-reported anxiety/depression, attention problems, and aggressive behavior later in life. *Archives of pediatrics & adolescent medicine*. 2008;162(4):330.
- 79. Hemmi MH, Wolke D, Schneider S. Associations between problems with crying, sleeping and/or feeding in infancy and long-term behavioural outcomes in childhood: a meta-analysis. *Archives of Disease in Childhood*. 2011;96(7):622-629.
- 80. Spoormaker VI, Montgomery P. Disturbed sleep in post-traumatic stress disorder: Secondary symptom or core feature? *Sleep Medicine Reviews*. 2008;12(3):169-184.
- 81. Harb GC, Cook JM, Gehrman PR, Gamble GM, Ross RJ. Post-traumatic stress disorder nightmares and sleep disturbance in Iraq war veterans: a feasible and promising treatment combination. *Journal of Aggression, Maltreatment & Trauma.* 2009;18(5):516-531.
- 82. Spilsbury JC. Sleep as a mediator in the pathway from violence-induced traumatic stress to poorer health and functioning: a review of the literature and proposed conceptual model. *Behavioral sleep medicine*. 2009;7(4):223-244.
- 83. Buysse D, Yu, L., Moul, D.E., Germain, A/. Stover, A., Dodds, N.E., Johnons, K.K., Shablesky-Cade, M.A., & Pilkonis, P. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. *Sleep.* 2010;33:1-12.
- 84. Delahaye J, Kovacs E, Sikora D, et al. The relationship between Health-Related Quality of Life and sleep problems in children with Autism Spectrum Disorders. *Research in Autism Spectrum Disorders*. 2014;8(3):292-303.
- 85. Jan JE, Owens JA, Weiss MD, et al. Sleep Hygiene for Children With Neurodevelopmental Disabilities. *Pediatrics*. 2008;122(6):1343-1350.


- 86. Owens JA. Classification and epidemiology of childhood sleep disorders. *Sleep Medicine Clinics*. 2007;2(3):353-361.
- 87. Adkins KW, Goldman SE, Fawkes D, et al. A pilot study of shoulder placement for actigraphy in children. *Behavioral sleep medicine*. 2012;10(2):138-147.
- 88. Goldman SE, McGrew S, Johnson K, Richdale A, Clemons T, Malow B. Sleep is associated with problem behaviors in children and adolescents with autism spectrum disorders. *Research in Autism Spectrum Disorders*. 2011;5:1223-1229.
- 89. Goldman SE, Richdale AL, Clemons T, Malow BA. Parental sleep concerns in autism spectrum disorders: Variations from childhood to adolescence. *Journal of Autism and Developmental Disorders*. 2012;42(4):531-538.
- 90. Krakowiak P, Goodlin-Jones B, Hertz- Piccioto I, Croen LA, Hansen RL. Sleep problems in children with autism spectrum disorders, developmental delays, and typical development: a population- based study. *Journal of Sleep Research*. 2008;17(2):197-206.
- 91. Polimeni MA, Richdale AL, Francis AJ. A survey of sleep problems in autism, asperger's disorder and typically developing children. *Journal of Intellectual Disability Research*. 2005;49(Pt 4):260-268.
- 92. Richdale AL, Prior MR. The sleep/wake rhythm in children with autism. *European Child and Adolescent Psychiatry*. 1995;4(3):175-186.
- 93. Richdale AL, Schreck KA. Sleep problems in autism spectrum disorders: Prevalence, nature, and possible biopsychosocial aetiologies. *Sleep Medicine Reviews*. 2009;13(6):403-411.
- 94. Souders MC, Mason TB, Valladares O, et al. Sleep behaviors and sleep quality in children with autism spectrum disorders. *Sleep*. 2009;32(12):1566-1578.
- 95. Turner KS, Johnson CR. Behavioral interventions to address sleep disturbances in children with autism spectrum disorders: A review. *Topics in Early Childhood Special Education*. 2012;33(3):144-152.
- 96. Vriend JL, Corkum PV, Moon EC, Smith IM. Behavioral interventions for sleep problems in children with autism spectrum disorders: current findings and future directions. *Journal of Pediatric Psychology*. 2011;36(9):1017-1029.
- 97. Johnson CR, Turner KS, Foldes E, Brooks MM, Kronk R, Wiggs L. Behavioral parent training to address sleep disturbances in young children with autism spectrum disorder: a pilot trial. *Sleep Medicine*. 2013;14(10):995-1004.
- 98. Allik H, Larsson JO, Smedje H. Sleep patterns of school-age children with asperger syndrome or high-functioning autism. *Journal of Autism and Developmental Disorders*. 2006;36(5):585-595.
- 99. Henderson JA, Barry TD, Bader SH, Jordan SS. The relation among sleep, routines, and externalizing behavior in children with an autism spectrum disorder. *Research in Autism Spectrum Disorders*. 2011;5(2):758-767.
- 100. Ibrahim SH, Voigt RG, Katusic SK, Weaver AL, Barbaresi WJ. Incidence of gastrointestinal symptoms in children with Autism: A population-based study. *Pediatrics*. 2009;124(2):680-686.
- 101. Reynolds AM, Malow BA. Sleep and autism spectrum disorders. *Pediatric Clinics of North America*. 2011;58(3):685-698.
- 102. Liu X, Hubbard JA, Fabes RA, Adam JB. Sleep disturbances and correlates of children with autism spectrum disorders. *Child Psychiatry & Human Development*. 2006;37(2):179-191.
- 103. Malow BA. Sleep disorders, epilepsy, and autism. *Mental Retardation and Developmental Disabilities Research Reviews.* 2004;10(2):122-125.
- 104. Melmed R, Schneider C, Fabes R, Phillips J, Reichelt K. Metabolic markers and gastrointestinal symptoms in children with autism and related disorders. *Journal of Pediatric Gastroenterology and Nutrition*. 2000;31:S31–32.
- 105. Valicenti-McDermott M, McVicar K, Rapin I, Wershil BK, Cohen H, Shinnar S. Frequency of gastrointestional symptoms in children with autistic spectrum disorders and association with family histry of autoimmune disease. *Journal of Developmental and Behavioiral Pediatrics*. 2006;27(2):S128-136.
- 106. Mazurek MOP, G.F. Sleep problems in childrne with autism spectrum disorder: Eamining the contributions of sensory over-responsivity and anxiety. *Sleep Medicine*. 2015;16:270-279.

- 107. Stores G, Wiggs L. Clinical services for sleep disorders. *Archives of Disease in Childhood*. 1998;79(6):495-497.
- 108. Malow BA, McGrew SG. Sleep disturbances and autism. Sleep Medicine Clinics. 2008;3(3):479-488.
- 109. Rossignol DA, Frye RE. Melatonin in autism spectrum disorders: a systematic review and metaanalysis. *Developmental Medicine & Child Neurology*. 2011;53(9):783-792.
- 110. Tordjman S, Anderson GM, Pichard N, Charbuy H, Touitou Y. Nocturnal excretion of 6-sulphatoxymelatonin in children and adolescents with autistic disorder. *Biological Psychiatry*. 2005;57(2):134-138.
- 111. Tordjman S, Anderson GM, Bellissant E, et al. Day and nighttime excretion of 6-sulphatoxymelatonin in adolescents and young adults with autistic disorder. *Psychoneuroendocrinology*. 2012;37(12):1990-1997
- 112. Gabriels RL, Cuccaro ML, Hill DE, Ivers BJ, Goldson E. Repetitive behaviors in autism: relationships with associated clinical features. *Research in Developmental Disabilities*. 2005;26(2):169-181.
- 113. Goldman SE, Surdyka K, Cuevas R, Adkins K, Wang L, Malow BA. Defining the sleep phenotype in children with autism. *Developmental neuropsychology*. 2009;34(5):560-573.
- 114. Malow BA, Marzec ML, McGrew SG, Wang L, Henderson LM, Stone WL. Characterizing sleep in children with autism spectrum disorders: a multidimensional approach. *Sleep.* 2006;29(12):1563-1571.
- 115. Schreck KA, Williams K, Smith AF. A comparison of eating behaviors between children with and without Autism. *Journal of Autism and Developmental Disorders*. 2004;34(4):433-438.
- 116. Mayes SD, Calhoun SL. Variables related to sleep problems in children with autism. *Research in Autism Spectrum Disorders*. 2009;3(4):931-941.
- 117. Mazurek MO, Sohl K. Sleep and behavioral problems in children with autism spectrum disorder. *Journal of Autism and Developmental Disorders*. 2016;46(6):1906-1915.
- 118. Richdale AL, Schreck KA. Sleep problems in autism spectrum disorders: prevalence, nature, & possible biopsychosocial aetiologies. *Sleep Med Rev.* 2009;13(6):403-411.
- 119. Hollway JA, Aman MG. Sleep correlates of pervasive developmental disorders: a review of the literature. *Research in Developmental Disabilities*. 2011;32(5):1399-1421.
- 120. Williams PG, Sears LL, Allard A. Sleep problems in children with autism. *Journal of Sleep Research*. 2004;13(3):265-268.
- 121. Lopez-Wagner MC, Hoffman CD, Sweeney DP, Hodge D, Gilliam JE. Sleep problems of parents of typically developing children and parents of children with autism. *The Journal of Genetic Psychology*. 2008;169(3):245-259.
- 122. Meltzer LJ. Brief report: sleep in parents of children with autism spectrum disorders. *Journal of Pediatric Psychology* 2008;33(4):380-386.
- 123. Meltzer LJ, Mindell JA. Relationship between child sleep disturbances and maternal sleep, mood, and parenting stress: a pilot study. *Journal of Family Psychology*. 2007;21(1):67-73.
- 124. Meltzer LJ. Factors associated with depressive symptoms in parents of children with autism spectrum disorders. *Research in Autism Spectrum Disorders*. 2011;5(1):361-367.
- 125. Doyen C, Mighiu D, Kaye K, et al. Melatonin in children with autistic spectrum disorders: recent and practical data. *European Child and Adolescent Psychiatry*. 2011;20(5):231-239.
- 126. Guénolé F, Godbout R, Nicolas A, Franco P, Claustrat B, Baleyte J-M. Melatonin for disordered sleep in individuals with autism spectrum disorders: Systematic review and discussion. *Sleep Medicine Reviews*. 2011;15(6):379-387.
- 127. Giannotti F, Cortesi F, Cerquiglini A, Bernabei P. An open-label study of controlled-release melatonin in treatment of sleep disorders in children with autism. *Journal of Autism and Developmental Disorders*. 2006;36(6):741-752.
- 128. Wasdell MB, Jan JE, Bomben MM, et al. A randomized, placebo-controlled trial of controlled release melatonin treatment of delayed sleep phase syndrome and impaired sleep maintenance in children with neurodevelopmental disabilities. *Journal of pineal research*. 2008;44(1):57-64.

- 129. Braam W, Didden R, Smits M, Curfs L. Melatonin treatment in individuals with intellectual disability and chronic insomnia: a randomized placebo- controlled study. *Journal of Intellectual Disability Research*. 2008;52(3):256-264.
- 130. Wright B, Sims D, Smart S, et al. Melatonin versus placebo in children with autism spectrum conditions and severe sleep problems not amenable to behaviour management strategies: a randomised controlled crossover trial. *Journal of Autism and Developmental Disorders*. 2011;41(2):175-184.
- 131. Harrington JW, Rosen L, Patrick PA. Parental perceptions and use of complementary and alternative medicine practices for children with autistic spectrum disorders in private practice. *Developmental and Behavioral Pediatrics*. 2006(27):S156-S161.
- 132. Andersen I, Kaczmarska J, McGrew S, Malow B. Melatonin for insomnia in children with autism spectrum disorders. *Journal of Child Neurology*. 2008;23(5):482-485.
- 133. Malow B, Adkins KW, McGrew SG, et al. Melatonin for sleep in children with autism: a controlled trial examining dose, tolerability, and outcomes. *Journal of Autism and Developmental Disorders*. 2012;42(8):1729-1737.
- 134. Mindell JA, Emslie G, Blumer J, et al. Pharmacologic Management of Insomnia in Children and Adolescents: Consensus Statement. *Pediatrics*. 2006;117(6):e1223-1232.
- 135. Malow BA, Byars K, Johnson K, et al. A practice pathway for the identification, evaluation, and management of insomnia in children and adolescents with autism spectrum disorders. *Pediatrics*. 2012;130 Suppl 2:S106-124.
- 136. Durand VM, Gernert-Dott P, Mapstone E. Treatment of sleep disorders in children with developmental disabilities. *Journal of the Association of Persons with Severe Handicap*. 1996;21:114–122.
- 137. Durand VM. Treating Sleep Terrors in Children with Autism. *Journal of Positive Behavior Interventions*. 2002;4(2):66-72.
- 138. Wolf MM, Risley T, Meese H. Application of operant conditioning procedures to the behavior problems of an autistic child. *Behavior Research and Therapy*. 1963;1(2):305-312.
- 139. Christodulu K, Durand VM. Reducing bedtime disturbance and night waking using positive bedtime routines and sleep restriction. *Focus on Autism and Other Developmental Disabilities*. 2004;19(3):130-139.
- 140. Durand VM, Christodulu K. Description of a sleep-restriction program to reduce bedtime disturbances and night waking. *Journal of Positive Behavior Interventions*. 2004;6(2):83-91.
- 141. Weiskop S, Richdale A, Matthews J. Behavioural treatment to reduce sleep problems in children with autism or fragile X syndrome. *Developmental Medicine & Child Neurology*. 2005;47(2):94-104.
- 142. Mindell JA, Kuhn B, Lewin DS, Meltzer LJ, Sadeh A. Behavioral treatment of bedtime problems and night wakings in infants and young children. *Sleep.* 2006;29(10):1263-1276.
- 143. Piazza CC, Fisher WW, Sherer M. Treatment of multiple sleep problems in children with developmental disabilities: faded bedtime with response cost versus bedtime scheduling. *Developmental Medicine & Child Neurology*. 1997;39(6):414-418.
- 144. Wiggs L, Stores G. Behavioural treatment for sleep problems in children with severe learning disabilities and challenging daytime behaviour: Effect on sleep patterns of mother and child. *Journal of Sleep Research*. 1998;7(2):119-126.
- 145. Weiskop S, Matthews J, Richdale A. Treatment of sleep problems in a 5-year-old boy with autism using behavioural principles. *Autism.* 2001;5(2):209-221.
- 146. Montgomery P, Stores G, Wiggs L. The relative efficacy of two brief treatments for sleep problems in young learning disabled (mentally retarded) children: a randomised controlled trial. *Archives of Disease in Childhood*. 2004;89(2):125-130.
- 147. Moon E, Corkum P, Smith I. Case study: A case-series evaluation of a behavioral sleep intervention for three children with autism and primary insomnia. *Journal of Pediatric Psychology*. 2010;36(1):47-54.
- 148. Aman MG, McDougle CJ, Scahill L, et al. Medication and parent training in children with pervasive developmental disorders and serious behavior problems: results from a randomized clinical trial. *Journal of American Academy of Child and Adolescent Psychiatry*. 2009;48(12):1143-1154.

Version 1.2: 7-12-2018

- 149. Scahill L, McDougle CJ, Aman MG, et al. Effects of Risperidone and parent training on adaptive functioning in children With pervasive developmental disorders and serious behavioral problems. *Journal of the American Academy of Child and Adolescent Psychiatry*. 2012;51(2):136-146.
- 150. Whittingham K, Sofronoff K, Sheffield J, Sanders M. Stepping Stones Triple P: an RCT of a parenting program with parents of a child diagnosed with an Autism Spectrum Disorder. *Journal of Abnormal Child Psychology*. 2009;37(4):469-480.
- 151. Aman MG, McDougle CJ, Scahill L, et al. Medication and parent training in children with pervasive developmental disorders and serious behavior problems: results from a randomized clinical trial. *Journal of American Academy of Child and Adolescent Psychiatry*. 2009;48(12):1143-1154.
- 152. Solomon M, Ono M, Timmer S, Goodlin-Jones B. The effectiveness of parent child interaction therapy for families of children on the autism spectrum. *Journal of Autism and Developmental Disorders*. 2008;38(9):1767-1776.
- 153. Tonge BJ, Brereton A, Kiomall M, MacKinnon A, King N, Rinehart N. Effects on parental mental health of an education and skills training program for parents of young children with autism: a randomized controlled trial. *Journal of American Academy of Child and Adolescent Psychiatry*. 2006;45(5):561-569.
- 154. Scahill L, Bearss K, Lecavalier L, et al. Effect of parent training on adaptive behavior in children with autism spectrum disorder and disruptive behavior: results of a randomized trial. *Journal of the American Academy of Child & Adolescent Psychiatry*. 2016;55(7):602-609.
- 155. Smith T, Scahill L, Dawson G, et al. Designing research studies on psychosocial interventions in autism. *Journal of Autism and Developmental Disorders*. 2007;37:354-366.
- 156. Cortesi F, Giannotti F, Sebastiani T, Panunzi S, Valente D. Controlled-release melatonin, singly and combined with cognitive behavioural therapy, for persistent insomnia in children with autism spectrum disorders: a randomized placebo-controlled trial. *Journal of Sleep Research*. 2012;21(6):700-709.
- 157. Malow B, Adkins K, Reynolds A, et al. Parent-Based Sleep Education for Children with Autism Spectrum Disorders. *Journal of Autism and Developmental Disorders*. 2014;44(1):216-228.
- 158. Dudding CC. Digital videoconferencing: Applications across the disciplines. *Communication Disorders Quarterly*. 2009;30(3):178-182.
- 159. Ingersoll B, Wainer AL, Berger NI, Pickard KE, Bonter N. Comparison of a self-directed and therapist-assisted telehealth parent-mediated intervention for children with ASD: A pilot RCT. *Journal of autism and developmental disorders*. 2016;46(7):2275-2284.
- 160. Vismara LA, McCormick C, Young GS, Nadhan A, Monlux K. Preliminary findings of a telehealth approach to parent training in autism. *Journal of Autism and Developmental Disorders*. 2013;43(12):2953-2969.
- 161. Wacker DP, Lee JF, Dalmau YCP, et al. Conducting functional communication training via telehealth to reduce the problem behavior of young children with autism. *Journal of developmental and physical disabilities*. 2013;25(1):35-48.
- 162. Suess AN, Wacker DP, Schwartz JE, Lustig N, Detrick J. Preliminary evidence on the use of telehealth in an outpatient behavior clinic. *Journal of applied behavior analysis*. 2016;49(3):686-692.
- 163. Pickard KE, Wainer AL, Bailey KM, Ingersoll BR. A mixed-method evaluation of the feasibility and acceptability of a telehealth-based parent-mediated intervention for children with autism spectrum disorder. *Autism.* 2016;20(7):845-855.
- 164. Johnson C, Foldes, E., Demand, A. Relationship between sleep of children with autism spectrum disorder and parental sleep quality. in preparation.
- 165. Sivertsen B, Posserud MB, Gillberg C, Lundervold AJ, Hysing M. Sleep problems in children with autism spectrum problems: a longitudinal population-based study. *Autism.* 2012;16(2):139-150.
- 166. Blunden S, Lushington K, Lorenzen B, Martin J, Kennedy D. Neuropsychological and psychosocial function in children with a history of snoring or behavioral sleep problems. *The Journal of Pediatrics*. 2005;146(6):780-786.

- 167. Ebert JCS, Drake AF. The impact of sleep-disordered breathing on cognition and behavior in children: A review and meta-synthesis of the literature. *Otolaryngology Head and Neck Surgery*. 2004;131(6):814.
- 168. Mindell JA, Emslie G, Blumer J, et al. Pharmacologic management of insomnia in children and adolescents: consensus statement. *Pediatrics*. 2006;117(6):e1223-1232.
- 169. Robins DL, Casagrande K, Barton M, Chen CM, Dumont-Mathieu T, Fein D. Validation of the Modified Checklist for Autism in Toddlers, revised with follow-up (M-CHAT-R/F). *Pediatrics*. 2014;133(1):37-45.
- 170. Rutter M, Bailey A, Lord C. *The Social Communication Questionnaire: Manual.* Torrance, CA: Western Psychological Services; 2003.
- 171. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)—a metadata-driven methodology and workflow process for providing translational research informatics support. *Journal of biomedical informatics*. 2009;42(2):377-381.
- 172. Guy W. Dosage Record and Treatment Emergent Symptoms Scale. *ECDEU Assessment Manual for Psychopharmacology (Revised)*. Rockville, MD.: US Department of Health, Education and Human Welfare publication (ADM); 1976:223-244.
- 173. Simonds J, Parraga H. Prevalence of sleep disorders and sleep behaviors in children and adolescents. *Journal of American Academy of Child and Adolescent Psychiatry*. 1982;21:383-388.
- 174. Spruyt K, Gozal D. Pediatric sleep questionnaire as diagnostic and epidemiological tools: A review of currently available instruments. *Sleep Medicine Reviews*. 2011;15:19-32.
- 175. Wiggs L, Stores G. Severe sleep disturbances and daytime challenging behavior in children with severe learning disabilities. *Journal of Intellectual Disability Research*. 1996;40:518-528.
- 176. Maas A, Didden R, Korzilius H, et al. Psychometric properties of a sleep questionnaire for use in individuals with intellectual disabilities. *Research in Developmental Disabilities*. 2011;32:2467-2479.
- 177. Scahill L, McCracken JT, King BH, et al. Extended-release guanfacine for hyperactivity in children with autism spectrum disorder. *American Journal of Psychiatry*. 2015;172(12):1197-1206.
- 178. Aman MG, Singh NN, Stewart AW, Field CJ. Psychometric characteristics of the Aberrant Behavior Checklist. *American Journal of Mental Deficiency*. 1985;89(5):492-502.
- 179. Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: A behavior rating scale for the assessment of treatment effects. *American Journal of Mental Deficiency*. 1985;89(5):485-491.
- 180. Shea S, Turgay A, Carroll A, et al. Risperidone in the treatment of disruptive behavioral symptoms in children with autistic and other pervasive developmental disorders. *Pediatrics*. 2004;114(5):e634-e641.
- 181. King BH, Hollander E, Sikich L, et al. Lack of efficacy of citalopram in children With autism spectrum disorders and high levels of repetitive behavior: citalopram ineffective in children with autism. *Archives of General Psychiatry*. 2009;66(6):583-590.
- 182. Network RUoPPRA. Risperidone in children with autism and serious behavioral problems. *New England Journal of Medicine*. 2002;347:314-321.
- 183. Network R. Risperidone treatment of autistic disorder: Longer term benefits and blinded discontinuation after six months. *American Journal of Psychiatry* 2005;162(7):1361-1369.
- 184. Aman MG, Singh NN. *Aberrant Behavior Checklist Manual, Second Edition*. East Aurora, NY: Slosson Educational Publications, Inc.; 2017.
- 185. Abidin R. Parenting Stress Index (3rd ed.). Lutz, FL: Psychological Assessment Resources; 1995.
- 186. Hassall R, Rose J, McDonald J. Parenting stress in mothers of children with an intellectual disability: the effects of parental cognitions in relation to child characteristics and family support. *Journal of Intellectual Disability Research*. 2005;49(6):405-418.
- 187. Montes G, Halterman JS. Characteristics of school-age children with autism. *Journal of Developmental and Behavioral Pediatrics*. 2006;27(5):379-385.
- 188. Wolery M, Garfinkle AN. Measures in intervention research with young children who have autism. *Journal of Autism and Developmental Disorders*. 2002;32(5):463.
- 189. Tomanik S, Harris GE, Hawkins J. The relationship between behaviours exhibited by children with autism and maternal stress. *Journal of intellectual & developmental disability.* 2004;29(1):16-26.


- 190. Postorino V, Gillespie S, Lecavalier L, et al. Clinical correlates of parenting stress in children with Autism Spectrum Disorder and serious behavioral problems. *Journal of Child and Adolescent Psychology*. In press.
- 191. Johnson C, Foldes E, DeMand A, Brooks M. Behavioral Parent Training to Address Feeding Problems in Children with Autism Spectrum Disorder: A Pilot Trial. *Journal of Developmental and Physical Disabilities*. 2015:1-17.
- 192. Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. *Journal of affective disorders*. 2009;114(1):163-173.
- 193. Gibaud-Wallson J, Wandersman LP. Development and utility of the Parenting Sense of Competence Scale. Paper presented at: American Psychological Association 1978; Toronto.
- 194. Gilmore L, Cuskelly M. Factor structure of the Parenting Sense of Competence scale using a normative sample. *Child: Care, health and development.* 2009;35(1):48-55.
- 195. Iadarola S, Levato L, Harrison B, et al. Teaching parents behavioral strategies for ASD: Effects on stress, strain and competence. *Journal of Autism and Developmental Disorders*. In press.
- 196. Buysse DJ, Reynolds III CF, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. *Psychiatry research*. 1989;28(2):193-213.
- 197. Johnson CR, Handen BL, Butter E, et al. Development of a parent training program for children with pervasive developmental disorders. *Behavioral Interventions*. 2007;22(3):201-221.
- 198. Bearss K, Johnson C, Handen B, Smith T, Scahill L. A pilot study of parent training in young children with autism spectrum disorders and disruptive behavior. *Journal of Autism and Developmental Disorders*. 2013;43(4):829-840.
- 199. Gurka MJ. Selecting the best linear mixed model under REML. *The American Statistician*. 2006;60(1):19-26.
- 200. Kenward MG, Roger JH. Small sample inference for fixed effects from restricted maximum likelihood. *Biometrics*. 1997:983-997.
- 201. Molenberghs G TH, Jansen I, Beunckens C, Kenward MG, Mallinckrodt C, Carroll RJ. Analyzing incomplete longitudinal clincal trial data. *Biostatiscis*. 2004;5(3):445-464.
- 202. Carpenter JR, Kenward MG. Missing data in randomised controlled trials-a practical guide. *Medical Statistics Unit, London School of Hygiene & Tropical Medicine: London School of Hygiene & Tropical Medicine.* 2007.
